CLINICAL TRIAL: NCT07014176
Title: A Multicenter, Randomized Trial Evaluating Dehydrated Human Placenta Tissue (dHPT) and Standard of Care Versus Standard of Care Alone in Nonhealing Diabetic Foot Ulcers
Brief Title: Nonhealing Diabetic Foot Ulcers Treated With Standard of Care (SOC) Alone or Standard of Care and Amnion-Intermediate-Chorion (AIC)
Acronym: ELITE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cellution Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CELLBIO-2025-001
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: DFU; Diabetic Ulcer; Foot Wound; Diabetic Foot Ulcer; Placenta
MeSH Terms: conditions — Diabetic Foot; Foot Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Interventions: Procedure: Standard of Care (SOC)
- AIC and Standard of Care (Experimental): Participants with a diabetic foot ulcer (DFU) will receive treatment with an Amnion-Intermediate-Chorion (AIC) sheet product, a dehydrated multilayer human placental tissue derived from donated human tissue, and weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Interventions: Other: Amnion-Intermediate-Chorion; Procedure: Standard of Care (SOC)

INTERVENTIONS:
Other: Amnion-Intermediate-Chorion — Dehydrated human placental multilayer allograft from derived donated human tissue. AIC contains amnion and chorion layers as well as basement membrane and trophoblast.
  Arms: AIC and Standard of Care
Procedure: Standard of Care (SOC) — Standard of care is to establish a clean, healthy wound bed and optimize the wound environment to have the best chance of healing the wound. This is achieved through wound cleansing, debridement, offloading and moisture balance.

SUMMARY:
The purpose of this study is to determine how well our dHPT (Dehydrated Human Placental Tissue) Product and Standard of Care work when compared to Standard of Care alone in achieving complete closure of diabetic foot.

DETAILED DESCRIPTION:
Chronic wounds affect a significant percentage of patients over their lifetime. For example, diabetic foot ulcers (DFU) are a major health complication that affect up to 15% of individuals with diabetes mellitus over their lifetime. The treatment of chronic wounds is extremely challenging as ulcers such as DFUs may not respond to standard of care (SOC) treatment and frequently become infected.

Advanced wound products like Dehydrated Human Placental Tissue (dHPTs) have become an important strategy in the treatment of these chronic wounds by trapping and binding the patients' own cells to rebuild the dermis layer of the skin to aid in healing.

This study will evaluate the clinical utility of Amnion-Intermediate-Chorion (AIC) in the closure of diabetic foot ulcers in subjects in comparison to Standard of Care treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible to participate in the study if the following conditions exist:

Inclusion Criteria:

1. 18 years of age or older.
2. Diagnosis of type 1 or 2 Diabetes mellitus.
3. Hemoglobin A1c (HbA1c) level is < 12% (108 mmol/mol).
4. Target ulcer with a surface area at randomization of 0.7 cm2 to 20.0 cm2 measured post debridement.
5. Target ulcer present for minimum of 4 weeks prior to screening visit.
6. Target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
7. Target ulcer must be Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the muscle provided it is below the medial aspect of the malleolus. The ulcer may not include exposed tendon or bone.
8. Affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the screening visit are acceptable:

   1. ABI ≥ 0.7 and ≤ 1.3;
   2. TBI ≥ 0.6;
   3. TCOM ≥ 40 mmHg;
   4. PVR: biphasic or triphasic.
9. Subject with two or more ulcers must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
10. Subject must consent to using the prescribed off-loading method for the duration of the study.
11. Subject must agree to attend study visits required by the protocol.
12. Subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

Subjects will be excluded from participation in the study if any of the following conditions exist:

1. Known life expectancy of < 6 months.
2. Target ulcer is not secondary to diabetes.
3. Target ulcer is infected or there is cellulitis in the surrounding skin.
4. Evidence of osteomyelitis complicating the target ulcer.
5. Infection in the target ulcer or a location that requires systemic antibiotic therapy.
6. Receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy is excluded.
7. Topical application of steroids to the ulcer surface within one month of screening.
8. Previous partial amputation on the affected foot if the resulting deformity impedes proper offloading of the target ulcer.
9. Surface area of the target ulcer has reduced in size by more than 20% in the 2 weeks prior to screening visit ("historical" run-in period). Photographic planimetry is not required for measurements taken during the historical run-in period (e.g. calculating surface area using length x width is acceptable).
10. Mini Nutritional Assessment (MNA) score of less than 17.
11. Acute Charcot foot or an inactive Charcot foot that impedes proper offloading of the target ulcer.
12. Women of childbearing potential (WOCBP) who are pregnant, considering becoming pregnant within the next 4 months, or are unwilling to use an appropriate form of contraception.
13. Currently require dialysis or planning to start dialysis.
14. Medical or psychological condition that, in the opinion of the investigator, may interfere with study assessments.
15. Treated with hyperbaric oxygen therapy or a dehydrated human placental tissue (dHTP) in the 30 days prior to screening visit.
16. Known sensitivity to ofloxacin, vancomycin, or amphotericin antibiotics.
17. Participation in a clinical trial involving treatment with an investigational product within the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of ulcers with complete wound closure | 1-12 weeks
  The percentage of DFU target ulcers achieving complete wound closure. Closure is defined as 100% re-epithelialization of the ulcer surface without detectable exudate.

SECONDARY OUTCOMES:
Time to complete closure for ulcer | 1-12 weeks
  Time to closure will be determined for the treatment group and compared to Standard of Care. Closure is defined by 100% re-epithelialization of the ulcer surface without detectable exudate.
Percentage of wound area change for target ulcer | 1-12 weeks
  Percentage wound area changes from week 1 to week 12 will be calculated weekly from measurements with digital photographic images and physical examination.
Changes to pain associated with the target ulcer | 1-12 weeks
  Change in pain in the target ulcer assessed using the Visual Analog Scale (VAS) from week 1 to week 12. VAS is a tool that uses a 0-10 (no to extreme pain) point scale to measure pain intensity.
Incidence of Adverse events | 1-12 weeks
  The incidence of adverse events will be evaluated weekly from the first study visit to wound healing and/or final visit.
Determine changes in Quality of Life | 1-12 weeks
  Changes in quality of life using both the Wound Quality of Life (wQOL) and Forgotten Wound Score (FWS) questionnaires that measure the health-related quality of life (HRQoL) of patients with chronic wounds. wQOL questionnaire is scored using a 5-point Likert scale, where 0 means "not at all" and 4 means "very much". Higher scores indicate greater impairment of quality of life. Higher the score indicates lower quality of life. [Time Frame: Visits 2, 5, 9, and 12/Final Visit]. FWS questionnaire measures 12 activities scored 0-4. Responses are summed and divided by the number of completed items. The mean value is then multiplied by 25 to obtain the total score of 0-100. Higher the score indicates lower quality of life. [Time Frame: Visits 2, 5, 9, and 12/Final Visit].

OTHER OUTCOMES:
Percentage of ulcers with complete wound closure for subjects 65 years or older | 1-12 weeks
  The percentage of DFU target ulcers in subjects 65 years or older achieving complete wound closure. Closure is defined by 100% re-epithelialization of the ulcer surface without detectable exudate.

CONTACTS AND LOCATIONS:
Overall Officials: Research Director, Study Director — Cellution Biologics
Locations (8):
- United States (8):
  - 005, Santa Rosa, California
  - 001, Jacksonville, Florida
  - 003, Chicago, Illinois
  - 007, Mooresville, North Carolina
  - 002, Rocky Mount, North Carolina
  - 008, Allentown, Pennsylvania
  - 004, Philadelphia, Pennsylvania
  - 006, Hilton Head Island, South Carolina

IPD SHARING:
Plan to Share IPD: No